CLINICAL TRIAL: NCT06820216
Title: The Analgesic Effects of Ultrasound Guided Recto-intercostal Facial Plane Block in Laparoscopic Hiatus Hernia Repair: A Double-Blind Randomized Controlled Study
Brief Title: Recto-intercostal Facial Plane Block in Laparoscopic Hiatus Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Marwa Ahmed Eloraby, lecturer of anesthesiology, surgical intensive care and pain medicine Tanta university, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 36264PR1064/1/25
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-01

CONDITIONS: Rectointercostal; Laparoscopic; Hiatus Hernia
Keywords: Ultrasound; Rectointercostal; Laparoscopic; Hiatus; Hernia
MeSH Terms: conditions — Hernia, Hiatal; Hernia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rectointercostal facial plane block group (Experimental): Patients will receive ultrasound-guided bilateral recto-intercostal facial plane block after induction of general anesthesia.
  Interventions: Drug: Rectointercostal facial plane block using bupivacaine 0.25%
- Control group (Other): Patients will receive general anesthesia without any block.
  Interventions: Other: No Intervention as a control

INTERVENTIONS:
Drug: Rectointercostal facial plane block using bupivacaine 0.25% — Ultrasound guided bilateral recto-intercostal facial plane block will be done after induction of general anesthesia using bupivacaine 0.25%. A linear ultrasound transducer Philips CX50 (5-14 MHz) will be placed 2-3 cm lateral and caudal to the xiphoid in the epigastric area. The rectus abdominis muscle and its insertion, 6th and 7th cartilage ribs will be visualized. The needle will be inserted between rectus abdominis muscle and the costal cartilages with an in-plane technique in a caudal-cranial way. Hydro-dissection will be performed with 5 ml saline for confirmation needle tip position, 20 ml of 0.25% bupivacaine will be injected, the same procedure will be then repeated with 20 ml 0.25% bupivacaine on the contra-lateral side (a total of 40 ml bilaterally).
  Arms: Rectointercostal facial plane block group
Other: No Intervention as a control — General anesthesia without performing any block.
  Arms: Control group

SUMMARY:
The aim of this study is to evaluate the perioperative analgesic and intraoperative hemodynamic effects of ultrasound-guided bilateral recto-intercostal fascial plane block in patients undergoing laparoscopic Hiatus hernia repair.

DETAILED DESCRIPTION:
Hiatus hernia is a prevalent condition in which the stomach or other abdominal organs protrude through the esophageal hiatus of the diaphragm into the thoracic cavity due to elevated pressure within the abdomen. Laparoscopic hernioplasty of hiatal hernia has been confirmed effective and safe in recent years and performed more due to its mini-invasive nature and intraperitoneal view and operating angle.

Although patients having laparoscopic hiatus hernia repair experience less pain than open surgery, postoperative pain can still be significant and lead to associated postoperative issues. These issues can include respiratory and other complications, delay in discharge and adverse effects from increasing requirements of systemic analgesia such as opioid. An important consideration in the potential multitude of problems associated with increased opioid use is respiratory depression, sedation, constipation and the propensity for vomiting. Postoperative vomiting can result in the repaired diaphragm enduring excessive pressure and subsequently early recurrence and failure of the procedure.

Recently, a novel block named "recto-intercostal fascial plane block" is performed between the recto abdominal muscle and costal cartilages of ribs 6-7 to block the anterior branches of the T6-T9 thoracic nerves, and laterally to the entire lower thorax. The investigators hypothesize that this block may provide perioperative analgesic benefits in patients undergoing Laparoscopic hiatus hernia repair under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years.
* American Society of Anesthesiology (ASA) physical status I-II.
* Both sexes.
* Type 1 hiatus hernia (sliding hiatus hernia) with gastro-esophageal reflux disease and scheduled for elective laparoscopic hiatus hernia repair under general anesthesia.

Exclusion Criteria:

* Patients with cardiovascular, pulmonary, or neurological diseases.
* History of chronic pain or Long-term or recent use of opioids.
* Coagulation disorders or infection at the block application area.
* History of allergy to local anesthetic drugs.
* History of previous abdominal surgery.
* Pregnancy.
* Patients with gastro-esophageal reflux disease complicated by high grade esophagitis, esophageal stenosis or bleeding, and aspiration pneumonia or asthma.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2025-02-17 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-08-21 (Actual)

PRIMARY OUTCOMES:
Total postoperative opioid consumption in the first 24 hours after surgery. | 24 hours after surgery.
  opioid dose (morphine 0.05 mg/kg) will be given to patients with pain score ≥ 4.

SECONDARY OUTCOMES:
Intraoperative fentanyl consumption. | End of surgery.
  Intravenous fentanyl bolus dosages of 1 μg/kg will be administered if intraoperative heart rate or mean arterial blood pressure elevated more than 20% of the baseline
Postoperative pain scores at post-anesthesia care unit arrival, 4 h, 8 h, 12 h, and 24 hour after surgery. | 24 hours after surgery.
  Numerical rating scale pain score (NRS) ranges from 0= no pain to 10= worst pain will be used to evaluate pain scores after surgery at rest and on movement from supine to sitting position.
Time to first postoperative opioid analgesic request. | 24 hours after surgery.
  opioid dose will be given to patients with pain score ≥ 4.
Side effects like postoperative nausea and vomiting, dysphagia and gas bloating after surgery | 24 hours after surgery.
  Any postoperative side effects will be reported.
Degree of patient satisfaction | 24 hour after surgery.
  The degree of patient satisfaction will be assessed before discharge by the Likert patient satisfaction scale: (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied; 5, extremely satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon reasonable request from the corresponding author.
Supporting Information: Study Protocol, SAP
Time Frame: After completion of the study.
Access Criteria: The data will be available upon reasonable request from the corresponding author.

REFERENCES:
- [Derived] Rehab OM, Bakr DM, El Malla DA, Helal RAEF, Morsy I, Eloraby M. The Analgesic Effects of Ultrasound-guided Recto-intercostal Fascial Plane Block in Laparoscopic Hiatus Hernia Repair: A Randomized Double-Blind Controlled Study. Anaesth Crit Care Pain Med. 2025 Dec 3:101724. doi: 10.1016/j.accpm.2025.101724. Online ahead of print. PMID 41349840